CLINICAL TRIAL: NCT05611307
Title: Detection of Late Subclinical Cardiovascular Disease in Testicular Cancer Survivors Exposed to Cisplatin-based Chemotherapy and Bone Marrow Transplant
Brief Title: Late Subclinical Cardiovascular Disease in Testicular Cancer Survivors
Status: Terminated | Type: Observational
Why Stopped: PI leaving Institution
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Suparna C. Clasen, Medical Director of Cardio-Oncology Director of Clinical Research Operations, Krannert Cardiovascular Research, Indiana University
Other Study IDs: 12751
Record Dates: First submitted 2022-10-21; First posted 2022-11-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Testicular Cancer; Survivorship; ASCVD; Coronary Artery Disease; Lipid Disorder; Hypogonadism, Male; Cisplatin Adverse Reaction; Bone Marrow Transplant Complications
MeSH Terms: conditions — Testicular Neoplasms; Coronary Artery Disease; Lipid Metabolism Disorders; Eunuchism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Surgical/Surveillance: TCS cured with surgical resection and surveillance (surgical/surveillance, Arm 1)
  Interventions: Diagnostic Test: Lipid profile; Diagnostic Test: Coronary artery assessment; Diagnostic Test: Hormone levels for hypogonadism
- Cisplatin-based chemotherapy (CBCT): TCS treat with one or more lines of cisplatin-based chemotherapy
  Interventions: Diagnostic Test: Lipid profile; Diagnostic Test: Coronary artery assessment; Diagnostic Test: Hormone levels for hypogonadism
- Cisplatin-based chemotherapy and Bone Marrow Transplant (CBCT/BMT): TCS treat with one or more lines of cisplatin-based chemotherapy, and who have undergone bone marrow transplant
  Interventions: Diagnostic Test: Lipid profile; Diagnostic Test: Coronary artery assessment; Diagnostic Test: Hormone levels for hypogonadism

INTERVENTIONS:
Diagnostic Test: Lipid profile — Advanced lipid profile
Diagnostic Test: Coronary artery assessment — Coronary artery assessment via CT scans
Diagnostic Test: Hormone levels for hypogonadism — Hormone levels for hypogonadism

SUMMARY:
Late subclinical cardiovascular disease in testicular cancer survivors exposed to cisplatin-based chemotherapy and bone marrow transplant

DETAILED DESCRIPTION:
Testicular cancer (TC) is diagnosed in young adult males between 18-39 years old. There are late (≥10 years after treatment) atherosclerotic cardiovascular disease (ASCVD) events after cisplatin-based chemotherapy (CBCT) treatment in testicular cancer survivors (TCS), along with heightened rates of hypertension, dyslipidemia, diabetes mellitus, and metabolic syndrome. Early detection of ASCVD to direct preventive measures in young TCS is an unmet need as these patients typically fall short of traditional 40-45-year age-cut offs for ASCVD screening. ASCVD risk will be evaluated in TCS ≥ 10 years after treatment in three groups: 1)TCS exposed to CBCT, 2)TCS exposed to CBCT and bone marrow transplant (BMT), and 3)TCS cured with surgical resection/surveillance. The focus will be on detecting subclinical atherosclerosis in TCS using blood lipid biomarkers and advanced cardiac CT imaging.

ELIGIBILITY:
Inclusion Criteria

* Patients >18 years of age
* Patients will be recruited only if cancer-free at clinical evaluation time.
* For the cases a confirmed TC diagnosis who received one or more cycles of CBCT-based chemotherapies (CBCT group, Arm 2)
* For the cases with a confirmed TC diagnosis who received one or more cycles of CBCT-based chemotherapies and underwent BMT for relapsed refractory disease (CBCT & BMT group, Arm 3).
* For the comparison cohort, biopsy-proven TC patients who had surgery for or surveillance of their testicular cancer and never received CBCTCBCT or BMT (surgical/surveillance, Arm 1)

Exclusion Criteria

* Prior known myocardial infarction (MI), atherosclerotic cardiovascular disease (ASCVD)
* Significant renal disease (GFR<40)
* Allergy to iodinated contrast
* Antecedent chemotherapy for another primary cancer.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Testicular Cancer Patients who are disease free more than 10 years after diagnosis and treatment
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Lipid profile | More than 10 years after testicular cancer diagnosis, At recruitment
  HDL, LDL, Tg, Cholesterol, Novel Lipid biomarkers using blood draws
Coronary plaque assessment | More than 10 years after testicular cancer diagnosis, At recruitment
  Coronary calcium score, coronary artery anatomy and plaque assessment using CT scans

SECONDARY OUTCOMES:
Hormone levels | More than 10 years after testicular cancer diagnosis, At recruitment
  Measurement of testosterone
Serum platinum | More than 10 years after testicular cancer diagnosis, At recruitment
  Measurement of residual serum platinum levels

CONTACTS AND LOCATIONS:
Overall Officials: Suparna C Clasen, MD MSCE, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No